CLINICAL TRIAL: NCT06413056
Title: Micafungin Versus Amphotercine B in Treatment of Invasive Fungal Infection In Preterm Neonates: A Randomized Control Trial
Brief Title: Micafungin Versus Amphotercine B in Treatment of Invasive Fungal Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ibrahim, Assistant Professor of Paediatrics, Ain Shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: micafungin in neonates
Record Dates: First submitted 2024-03-11; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neonatal Infection; Invasive Fungal Infections
Keywords: preterm; neonate; invasive fungal infection; micafungin
MeSH Terms: conditions — Invasive Fungal Infections; Premature Birth | interventions — Micafungin; Amphotericin B

STUDY DESIGN:
Intervention Model Description: Primary aim; to study the effectiveness of micafungin in treatment of fungal infection in preterm neonates.
  Secondary aim; to test the safety of micafungin in treatment of fungal infection in preterm neonates.
  Tertiary aim; to compare the effectiveness and safety of micafungin versus amphotericin B in treatment of invasive fungal infection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized controlled, Double Blinded Clinical Trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- micafungin group (Experimental): Preterm neonate with fungal infection provened by fungal culture and who received fluconazole for at least one week will be divided into two groups. Will receive micafungin at a dose of 8 mg/kg/day for 14 day (Auriti et al., 2016).
  Interventions: Drug: Micafungin
- amphotericin B group (Active Comparator): Preterm neonate with fungal infection provened by fungal culture and who received fluconazole for at least one week will be divided into two groups. Will receive amphotericin B at a dose of 1 mg /kg/day for 14 days (chen et al.,2019).
  Interventions: Drug: Amphotericin B

INTERVENTIONS:
Drug: Micafungin — Preterm neonate with fungal infection provened by fungal culture and who received fluconazole for at least one week will be divided into two groups. Will receive either micafungin or amphotericin B
  Arms: micafungin group
Drug: Amphotericin B — Preterm neonate with fungal infection provened by fungal culture and who received fluconazole for at least one week will be divided into two groups.
  Arms: amphotericin B group

SUMMARY:
The incidence of fungal infection has increased dramatically over the past few decades.This is due to increase in survival rates of preterm neonates, advances in medical technology and drug therapy, broad spectrum antibiotics and parenteral nutrition . The resistance to antifungal agents has increased. This study will assess the efficacy of micafungin versus amphotericin B in neonates with positive fungal culture.

DETAILED DESCRIPTION:
Neonatal candidiasis is associated with significant mortality and morbidity and high rates of neuro-developmental impairment on follow up Prevalence of invasive fungal infection (IFI) has increased in neonates during the last two decades due to increased survival rate even in the extremely premature neonates. Candida albicans and Candida parapsilosis are responsible for the majority of candidiasis in the neonatal intensive care unit (NICU) According to the European Society for Clinical Microbiology and Infectious Diseases (ESCMID)guidelines published in 2012, Micafungin, amphotericin B deoxycholate, and fluconazole are recommended as first line treatment of invasive candidiasis in neonates Currently, fluconazole and micafungin are among the most frequently used antifungal agents for the treatment of neonatal invasive candidiasis High dose of micafungin (8 to 15 mg/kg/day) can be used with neonates and infant with invasive candidiasis In this study we will explore the effectiveness and safety of micafungin for treatment of candidiasis after fluconazole for preterm neonates with invasive fungal infection and to compare it with amphotericin B.

ELIGIBILITY:
Inclusion Criteria:

* Patient less than 36 weeks gestational age
* started fluconazole either prophylactic or therapeutic dose
* and blood culture is positive for fungal infection.

Exclusion Criteria:

* Any neonate with hepatic dysfunction for any cause (hepatitis or hepatic failure), or with elevation in AST, ALT, alkhaline phosphatase
* Any neonate hypertensive, neutropenic, thrombocytopenic
* Any neonate with elevated renal function
* Any neonate with arrythmia

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
resolution of fungal infection | 14 days
  negative blood culture

SECONDARY OUTCOMES:
complication | one month
  drug complications
morbidity | one month
  hospital stay
mortality | one month
  death

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim MJA, Mohammed Fathy MS, Ghobrial MAT, Mohamed MH. Micafungin versus Amphotericin B in treatment of invasive fungal infection in preterm neonates: a randomized control trial. Ital J Pediatr. 2025 Feb 27;51(1):61. doi: 10.1186/s13052-025-01852-9. PMID 40016807